CLINICAL TRIAL: NCT04566887
Title: A Phase II Study of Acalabrutinib in Combination With R-CHOP Chemotherapy in Previously Untreated Mantle Cell Lymphoma
Brief Title: Acalabrutinib With R-CHOP in Previously Untreated Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-109; 20-5858 (Other: UHN)
Record Dates: First submitted 2020-09-15; First posted 2020-09-28 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — acalabrutinib; R-CHOP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (Experimental): Acalabrutinib 100mg twice per day orally with standard of care R-CHOP chemotherapy by IV every 21 days for a maximum of six cycles. After 6 cycle of R-CHOP and study drug eligible participants will undergo ASCT.
  Interventions: Drug: Acalabrutinib; Drug: R-CHOP chemotherapy
- Cohort B (Experimental): Acalabrutinib 100mg twice per day orally with standard of care R-CHOP chemotherapy by IV every 21 days for a maximum of six cycles.
  Interventions: Drug: Acalabrutinib; Drug: R-CHOP chemotherapy

INTERVENTIONS:
Drug: Acalabrutinib — Administered as 100mg tablets.
Drug: R-CHOP chemotherapy — R-CHOP chemotherapy

SUMMARY:
This is a multicenter, open-label, non-randomized, phase II clinical trial conducted in Canada. The purpose of the study is to determine the remission rate of acalabrutinib in combination with R-CHOP in patients with previously untreated mantle cell lymphoma prior to autologous stem cell transplantation. This study is composed of 2 cohorts, A and B. In Cohort A all patients will receive six cycles of R-CHOP chemotherapy together with continuous acalabrutinib at the standard dose twice per day orally. All patients will undergo response assessment at the end of six cycles of R-CHOP + acalabrutinib with CT scan, PET/CT scan, and bone marrow biopsy. Responding patients will proceed with stem cell mobilization, apheresis, and processing. Following ASCT, patients will receive standard maintenance rituximab every 3 months for 2 years. Enrollment for Cohort A component of the study has been completed. Cohort B, involves using acalabrutinib with R-CHOP (same as Group A) but without an autologous stem cell transplant (ASCT) as part of the regimen. The study doctors hope to evaluate how participants respond to the treatment in terms of the time between treatment initiation and time when stable disease is achieved. The enrollment for cohort B is currently ongoing.

ELIGIBILITY:
Cohort A:

Inclusion Criteria Eligible subjects will be considered for inclusion in Cohort A of this study if they meet all of the following criteria:

1. Men and women greater than or equal to 18 years of age deemed eligible for treatment with Full dose RCHOP and ASCT by the qualified investigator.
2. Histologic diagnosis of MCL according to the World Health Organization classification [Swerdlow, Blood 2016].
3. Previously untreated MCL with the following exceptions: (a) prior radiotherapy for localized disease, (b) up to 7 days of corticosteroids (prednisone 100mg/day equivalent), (c) up to one dose of single-agent chemotherapy (for example, cyclophosphamide), (d) up to one cycle of R-CHOP if last R-CHOP is between 21 days and 2 months from start of RCHOP+acalabrutinib or up to one cycle ofbendamustine-rituximab (BR) if BR is between 28 days and 2 months from start of RCHOP+acalabrutinib. Patients with exceptions (c) and (d) are eligible as long as all other eligibility criteria are met AND at least a CT scan and bone marrow biopsy were performed prior to chemotherapy.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
5. Presence of at least one radiologically measurable nodal or extranodal mass. A measurable nodal mass must have a longest diameter ≥1.5 cm. A measurable extranodal mass should have a longest diameter ≥1.0 cm.[Cheson, JCO 2014]
6. Women of childbearing potential (WOCBP) who are sexually active must use highly effective methods of contraception during treatment and up to 12 months after the last dose of rituximab or R-CHOP, or 2 days after the last dose of acalabrutinib, whichever is last administered. Examples of highly effective contraceptive methods include an agreement to remain abstinent (ie, refrain from heterosexual intercourse), bilateral tubal ligation, male sterilization, established proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. Men who are sexually active must use highly effective methods of contraception during treatment and up to 6 months after the last dose of rituximab or R-CHOP, or 2 days after the last dose of acalabrutinib, whichever is last administered. Men require an agreement to remain abstinent (ie, refrain from heterosexual intercourse) or use a condom, and an agreement to refrain from donating sperm. Periodic abstinence and withdrawal are not acceptable methods of contraception. Fertility preservation options should be discussed.
7. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty.
8. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information.

Exclusion Criteria:

Subjects will be ineligible for Cohort A of this study if they meet any of the following criteria:

1. Secondary central nervous system involvement.
2. Prior exposure to a BCR inhibitor (eg, BTK inhibitors, phosphoinositide-3 kinase (PI3K), or Syk inhibitors) or BCL-2 inhibitor.
3. Prior malignancy (or any other malignancy requiring active treatment), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical or prostate cancer, or other cancer from which the subject has been disease free for ≥ 3 years or which will not limit survival to < 5 years. Subjects receiving adjuvant hormonal therapy for early breast or prostate cancer are eligible.
4. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification. Subjects with controlled, asymptomatic atrial fibrillation during screening can enroll on study.
5. Difficulty with or unable to swallow oral medication, or conditions significantly affecting gastrointestinal function that would limit absorption of oral medication.
6. Known history of infection with HIV or any significant active infection (eg, bacterial, viral or fungal), including suspected or confirmed progressive multifocal leukoencephalopathy.
7. Known history of drug-specific hypersensitivity or anaphylaxis to study drugs (acalabrutinib and individual components of R-CHOP), including active product or excipient components.
8. Active bleeding or history of bleeding diathesis (eg, hemophilia or von Willebrand disease).
9. Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura).
10. Requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducer which cannot be modified as described in Sections 3.8.2 and 3.9.2, and/or the dose of acalabrutinib cannot be modified as described in these sections.
11. Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (eg, warfarin).
12. Requires treatment with proton pump inhibitors (eg, omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study.
13. History of significant cerebrovascular disease/event, including stroke or intracranial hemorrhage, within 6 months before the first dose of study drug.
14. Major surgical procedure within 4 weeks of first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
15. Received a live virus vaccination within 28 days of first dose of R-CHOP + acalabrutinib.
16. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (antiHBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR) result before enrolment and must be willing to undergo PCR testing during the study. Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded.Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded. Subjects with a history of Hepatitis C who received antiviral treatment are eligible as long as PCR is negative.
17. ANC <1.0 x109/L (subjects with bone marrow involvement by lymphoma are eligible regardless of ANC)
18. Platelets <50 x109/L (subjects with bone marrow involvement by lymphoma are eligible regardless of platelet count)
19. Total serum bilirubin ≥1.5 times the upper limit of normal, unless directly attributable to Gilbert's syndrome (or >3 times for documented hepatic involvement by lymphoma), AST and ALT >3 times the upper limit of normal (or >5 times for documented hepatic involvement by lymphoma)
20. Creatinine clearance <30 mL/min.
21. PT/INR >2 times the upper limit of normal in the absence of anticoagulants and/or PTT >2 times the upper limit of normal in the absence of anticoagulants.
22. Breastfeeding or pregnant. WOCBP must have a serum and/or urine pregnancy test done a maximum of 7 days prior to treatment initiation and a negative result must be documented prior to recruitment.
23. Concurrent participation in another therapeutic clinical trial.
24. Evidence of disease (such as severe or uncontrolled systemic diseases, including uncontrolled hypertension and renal transplant) that, in the investigator's opinion, make it undesirable for the patient to participate in the study or that would jeopardize compliance with the protocol.
25. Received any investigational drug within 30 days or 5 half-lives (whichever is shorter) before first dose of study drug.
26. Current life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the subject's safety or put the study at risk.

Cohort B:

Inclusion Criteria:

Eligible subjects will be considered for inclusion in Cohort B of this study if they meet all of the following criteria:

1. Men and women 18-70 years of age deemed eligible for treatment with full dose RCHOP by the qualified investigator.
2. Histologic diagnosis of MCL according to the World Health Organization classification [Swerdlow, Blood 2016].
3. Previously untreated MCL with the following exceptions: (a) prior radiotherapy for localized disease, (b) up to 7 days of corticosteroids (prednisone 100mg/day equivalent), (c) up to one dose of single-agent chemotherapy (for example, cyclophosphamide), (d) up to one cycle of R-CHOP if last R-CHOP is between 21 days and 2 months from start of R-CHOP+acalabrutinib. Other chemotherapy regimens (for example, bendamustine and rituximab) are not allowed. Patients with exceptions (c) and (d) are eligible as long as all other eligibility criteria are met AND at least a CT scan and bone marrow biopsy were performed prior to chemotherapy.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
5. Presence of at least one radiologically measurable nodal or extranodal mass. A measurable nodal mass must have a longest diameter ≥1.5 cm. A measurable extranodal mass should have a longest diameter ≥1.0 cm.[Cheson, JCO 2014]
6. Women of childbearing potential (WOCBP) who are sexually active must use highly effective methods of contraception during treatment and up to 12 months after the last dose of rituximab or R-CHOP, or 2 days after the last dose of acalabrutinib, whichever is last administered. Examples of highly effective contraceptive methods include an agreement to remain abstinent (ie, refrain from heterosexual intercourse), bilateral tubal ligation, male sterilization, established proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. Men who are sexually active must use highly effective methods of contraception during treatment and up to 6 months after the last dose of rituximab or R-CHOP, or 2 days after the last dose of acalabrutinib, whichever is last administered. Men require an agreement to remain abstinent (ie, refrain from heterosexual intercourse) or use a condom, and an agreement to refrain from donating sperm. Periodic abstinence and withdrawal are not acceptable methods of contraception. Fertility preservation options should be discussed.
7. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules or tablets without difficulty.
8. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information

Exclusion Criteria:

Subjects will be ineligible for Cohort B of this study if they meet any of the following criteria:

1. Secondary central nervous system involvement.
2. Prior exposure to a BCR inhibitor (eg, BTK inhibitors, phosphoinositide-3 kinase (PI3K), or Syk inhibitors) or BCL-2 inhibitor.
3. Prior malignancy (or any other malignancy requiring active treatment), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical or prostate cancer, or other cancer from which the subject has been disease free for ≥ 3 years or which will not limit survival to < 5 years. Subjects receiving adjuvant hormonal therapy for early breast or prostate cancer are eligible.
4. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification. Subjects with controlled, asymptomatic atrial fibrillation during screening can enroll on study.
5. Difficulty with or unable to swallow oral medication, or conditions significantly affecting gastrointestinal function that would limit absorption of oral medication.
6. Known history of infection with HIV or any significant active infection (eg, bacterial, viral or fungal), including suspected or confirmed progressive multifocal leukoencephalopathy.
7. Known history of drug-specific hypersensitivity or anaphylaxis to study drugs (acalabrutinib and individual components of R-CHOP), including active product or excipient components.
8. Active bleeding or history of bleeding diathesis (eg, hemophilia or von Willebrand disease).
9. Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura).
10. Requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducer which cannot be modified as described in Sections 3.8.2 and 3.9.2, and/or the dose of acalabrutinib cannot be modified as described in these sections.
11. Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (eg, warfarin).
12. History of significant cerebrovascular disease/event, including stroke or intracranial hemorrhage, within 6 months before the first dose of study drug.
13. Major surgical procedure within 4 weeks of first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
14. Received a live virus vaccination within 28 days of first dose of R-CHOP + acalabrutinib.
15. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR) result before enrolment and must be willing to undergo PCR testing during the study. Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded. Subjects with a history of Hepatitis C who received antiviral treatment are eligible as long as PCR is negative.
16. ANC <1.0 x109/L (subjects with bone marrow involvement by lymphoma are eligible regardless of ANC)
17. Platelets <50 x109/L (subjects with bone marrow involvement by lymphoma are eligible regardless of platelet count)
18. Total serum bilirubin ≥1.5 times the upper limit of normal, unless directly attributable to Gilbert's syndrome (or >3 times for documented hepatic involvement by lymphoma), AST and ALT >3 times the upper limit of normal (or >5 times for documented hepatic involvement by lymphoma)
19. Creatinine clearance <30 mL/min.
20. PT/INR >2 times the upper limit of normal in the absence of anticoagulants and/or PTT >2 times the upper limit of normal in the absence of anticoagulants.
21. Breastfeeding or pregnant. WOCBP must have a serum and/or urine pregnancy test done a maximum of 7 days prior to treatment initiation and a negative result must be documented prior to recruitment.
22. Concurrent participation in another therapeutic clinical trial.
23. Evidence of disease (such as severe or uncontrolled systemic diseases, including uncontrolled hypertension and renal transplant) that, in the investigator's opinion, make it undesirable for the patient to participate in the study or that would jeopardize compliance with the protocol.
24. Received any investigational drug within 30 days or 5 half-lives (whichever is shorter) before first dose of study drug.
25. Current life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the subject's safety or put the study at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2032-04-30 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate by PET/CT scan using Lugano Classification for Malignant Lymphoma - Cohort A | 1-2 weeks after completing six cycles (21 days) of R-CHOP + acalabrutinib.
To evaluate FFS in patients receiving acalabrutinib + R-CHOP followed by 2 years of maintenance acalabrutinib + rituximab - Cohort B | 2-year failure-free survival (FFS), defined as time from treatment initiation to stable disease after at least 4 cycles of induction, relapse/progression at any time, or death from any cause

SECONDARY OUTCOMES:
Adverse events of acalabrutinib and R-CHOP by using CTCAE version 5.0 | Baseline through end of study treatment (up to 18 weeks)
Measures of efficacy by using the RECIL 2017 criteria. | Baseline to end of study (up to 2 years)
Rate of minimal residual disease negativity (MRD) prior to transplant by flow cytometry | Up to 18 weeks
Event-free in patients who discontinue acalabrutinib at the point of MRD negativity prior to transplant by flow cytometry | Baseline to end of study (up to 2 years)
Changes in scores of partient reported outcomes (PRO) as measured by FACT-Lym | Baseline to end of study (up to 2 years)
  Composed of the FACT-G plus the 15-item Lymphoma Subscale (LymS).
Overall survival in patients who discontinue acalabrutinib at the point of MRD negativity | Baseline to end of study (up to 2 years)
Changes in scores of partient reported outcomes (PRO) as measured by FACT-Cog | Baseline to end of study (up to 2 years)
  Participants rated their cognitive function on a scale of 0 to 4 where 0 was never and 4 was several times a day.
Changes in scores of partient reported outcomes (PRO) as measured by EORTC QLQ-C30 | Baseline to end of study (up to 2 years)
  Participants rated their quality of life on a scale of 1 to 4 where 1 was not at all and 4 was very much.
To evaluate event-free and overall survival in patients who achieve MRD negativity | Baseline to end of study (up to 2 years)

OTHER OUTCOMES:
To explore the use of tumor-specific circulating DNA in plasma/serum as a non-invasive diagnostic and prognostic tool, with paired diagnostic tissue material, through treatment of MCL and at follow-up | Baseline to end of study (up to 2 years)
To explore the performance of the MCL proliferation signature, assessed using the MCL35 assay, in patients receiving BTK inhibition in combination with chemoimmunotherapy. | Baseline to end of study (up to 2 years)
To explore the use of microRNAs in plasma serum through treatment of MCL and at follow-up. | Baseline to end of study (up to 2 years)

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - BC Cancer Agency, Vancouver, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Centre Hospitalier Universitaire de Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Undecided